CLINICAL TRIAL: NCT02829268
Title: A Phase 1b/2a Trial of Dantrolene Sodium in Pediatric and Adult Patients With Wolfram Syndrome
Brief Title: A Clinical Trial of Dantrolene Sodium in Pediatric and Adult Patients With Wolfram Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201607006; R21DK113487 (NIH)
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Wolfram Syndrome; Diabetes Mellitus; Optic Nerve Atrophy; Ataxia
Keywords: Wolfram syndrome; Diabetes Mellitus; Optic Nerve Atrophy; Ataxia; Endoplasmic Reticulum Stress
MeSH Terms: conditions — Wolfram Syndrome; Diabetes Mellitus; Optic Atrophy; Ataxia | interventions — Dantrolene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pediatric (Experimental): Pediatric patients treated with dantrolene sodium
  Interventions: Drug: dantrolene sodium
- Adult (Experimental): Adult patients treated with dantrolene sodium
  Interventions: Drug: dantrolene sodium

INTERVENTIONS:
Drug: dantrolene sodium — The purpose of this study is to assess the safety and tolerability of dantrolene sodium in patients with Wolfram syndrome. In addition, we will assess the efficacy of dantrolene sodium on the cardinal manifestations of Wolfram syndrome, including visual acuity, remaining beta cell functions, and neurological functions.
  There is a screening period up to 56 days, a 6-month treatment period with an optional extension phase up to 24 months, and a 4-week safety follow-up period. Study assessments include medical & medication history, physical exams, neurological exams, eye exams, endocrine exams, vital signs, height, weight, electrocardiograms, blood and urine tests, pregnancy test if applicable, and questionnaires.
  Other Names: dantrolene

SUMMARY:
Wolfram syndrome is a rare genetic disorder characterized by juvenile-onset diabetes mellitus, diabetes insipidus, optic nerve atrophy, hearing loss, and neurodegeneration. The purpose of this study is to assess the safety and tolerability of dantrolene sodium in patients with Wolfram syndrome. In addition, we will assess the efficacy of dantrolene sodium on the cardinal manifestations of Wolfram syndrome, including visual acuity, remaining beta cell functions, and neurological functions.

There is a screening period up to 56 days, a 6-month treatment period with an optional extension phase up to 24 months, and a 4-week safety follow-up period. Study assessments include medical & medication history, physical exams, neurological exams, eye exams, endocrine exams, vital signs, height, weight, electrocardiograms, blood and urine tests, pregnancy test if applicable, and questionnaires.

DETAILED DESCRIPTION:
The Primary Objective of this study is:

To assess the safety and tolerability of dantrolene sodium administered orally at upper end of therapeutic dose range for 6 months in patients with Wolfram syndrome with an optional extension phase up to 24 months. Patients who express the wish to continue in the optional extension phase on dantrolene sodium will be offered this possibility.

The Secondary Objectives of this study are:

* Determine the effect of dantrolene sodium on remaining beta cell functions using a mixed-meal tolerance test and monitoring base-line C-peptide levels, blood glucose levels, proinsulin/C-peptide ratios, hemoglobin A1c levels, and urine glucose levels.
* To determine the efficacy of dantrolene sodium on visual acuity (LogMar scores)
* To determine the efficacy of dantrolene sodium on visual functions using Visual Functioning Questionnaire - 25.
* To evaluate the efficacy of dantrolene sodium on neurological functions using the Wolfram Unified Rating Scale (WURS) and standard neurological assessments.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrolment:

1. The patient has a definitive diagnosis of Wolfram syndrome, as determined by the following:

   a. Documented functionally relevant recessive mutations on both alleles of the WFS1 gene or dominant mutation on one allele of the WFS1 gene based on historical test results (if available) or from a qualified laboratory at screening.
2. The patient is at least 5 years of age (biological age) at the time of written informed consent.
3. The patient, patient's parent(s), or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient. The guardians' consent and patient's assent, as relevant, must be obtained.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study:

1. The patient has clinically significant non-Wolfram related CNS involvement which is judged by the investigator to be likely to interfere with the accurate administration and interpretation of protocol assessments.
2. The patient has a known defect in oxidative phosphorylation (such as a confirmed mitochondrial myopathy)
3. The patient has abnormal liver function (defined as serum transaminases more than twice the upper limit of normal for the reference laboratory)
4. The patient has a significant medical or psychiatric co-morbidity that might affect study data or confound the integrity of study results.
5. The patient has received treatment with any investigational drug within the 30 days prior to study entry.
6. The patient has received blood product transfusions within 90 days prior to screening.
7. The patient is unable to comply with the protocol, (e.g. has a clinically relevant medical condition making implementation of the protocol difficult, unstable social situation, known clinically significant psychiatric/behavioural instability, is unable to return for safety evaluations, or is otherwise unlikely to complete the study), as determined by the Investigator.
8. The patient has a known history of central apnea and/or ventilation requirements.
9. The patient has a known history of chronic obstructive pulmonary disease, pleural effusion, and/or myocardial disease.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fumihiko Urano, MD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We publish aggregated data in a scientific journal.

REFERENCES:
- [Background] Urano F. Wolfram Syndrome: Diagnosis, Management, and Treatment. Curr Diab Rep. 2016 Jan;16(1):6. doi: 10.1007/s11892-015-0702-6. PMID 26742931
- [Result] Abreu D, Stone SI, Pearson TS, Bucelli RC, Simpson AN, Hurst S, Brown CM, Kries K, Onwumere C, Gu H, Hoekel J, Tychsen L, Van Stavern GP, White NH, Marshall BA, Hershey T, Urano F. A phase Ib/IIa clinical trial of dantrolene sodium in patients with Wolfram syndrome. JCI Insight. 2021 Aug 9;6(15):e145188. doi: 10.1172/jci.insight.145188. PMID 34185708
- See also: Wolfram Syndrome Center — https://wolframsyndrome.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric: Pediatric patients treated with dantrolene sodium
  dantrolene sodium: The purpose of this study is to assess the safety and tolerability of dantrolene sodium in patients with Wolfram syndrome. In addition, we will assess the efficacy of dantrolene sodium on the cardinal manifestations of Wolfram syndrome, including visual acuity, remaining beta cell functions, and neurological functions.
  There is a screening period up to 56 days, a 6-month treatment period with an optional extension phase up to 24 months, and a 4-week safety follow-up period. Study assessments include medical & medication history, physical exams, neurological exams, eye exams, endocrine exams, vital signs, height, weight, electrocardiograms, blood and urine tests, pregnancy test if applicable, and questionnaires.
- Adult: Adult patients treated with dantrolene sodium
  dantrolene sodium: The purpose of this study is to assess the safety and tolerability of dantrolene sodium in patients with Wolfram syndrome. In addition, we will assess the efficacy of dantrolene sodium on the cardinal manifestations of Wolfram syndrome, including visual acuity, remaining beta cell functions, and neurological functions.
  There is a screening period up to 56 days, a 6-month treatment period with an optional extension phase up to 24 months, and a 4-week safety follow-up period. Study assessments include medical & medication history, physical exams, neurological exams, eye exams, endocrine exams, vital signs, height, weight, electrocardiograms, blood and urine tests, pregnancy test if applicable, and questionnaires.
Period: Overall Study
Arm/Group | Pediatric | Adult
Started | 8 | 13
Completed | 8 | 11
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric | Adult | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 0 | 8
  Between 18 and 65 years | 0 | 11 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 13 [6 to 17] | 23 [18 to 32] | 18 [6 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19
Abnormal liver function test results [Count of Participants; unit: Participants] — The investigators perform liver function tests to check the levels of certain enzymes and proteins in participants' blood. Levels that are higher or lower than normal can indicate liver problems. The liver function tests include:
  Alanine transaminase (ALT), Aspartate transaminase (AST), Alkaline Phosphatase (AP), and bilirubin.
  Participants | 0 | 0 | 0
C-peptide levels in participants during the oral mixed meal tolerance test [Mean (Standard Deviation); unit: ng/mL] — The investigators track C-peptide levels in participants' blood throughout the oral mixed meal tolerance test. Blood samples for glucose and C-peptide measurement are taken at two points: at the start (fasting, time 0) and 30 minutes after the Boost. The difference in C-peptide levels between these two time points is calculated by subtracting the value at 0 minutes from the value at 30 minutes.
  ng/mL | 0.34 (0.07) | 0.19 (0.05) | 0.25 (0.04)
Visual Functioning in participants assessed by Visual Functioning Questionnaire-25 [Mean (Standard Deviation); unit: units on a scale] — The Visual Functioning Questionnaire-25 (VFQ-25) is divided into several subdomains. There are a total of 11 subdomains in the VFQ-25. To calculate the total score on the VFQ-25, we follow these steps:1. Calculate Subdomain Scores, 2. Weighted Sum 3. Calculate Total Score.
  VFQ-25 provides scores that range from 0 to 100. The total score represents the overall impact of visual functioning on the individual's quality of life, with higher scores indicating better quality of life and less impact from vision problems.
  units on a scale | 68 (2.3) | 74.3 (1.3) | 68.8 (3.1)
Best-corrected visual acuity in participants measured by LogMar Score [Mean (Standard Deviation); unit: LogMAR] — Best-corrected visual acuity is assessed using the Snellen optotype and then converted into LogMar Scores (Minimum: -0.30, Maximum: 3.0). A higher LogMar score signifies poorer vision.
  LogMAR | 0.6 (0.2) | 0.8 (0.2) | 0.7 (0.2)
Neurological Functions in participants assessed by the Wolfram Unified Rating Scale (WURS) [Mean (Standard Deviation); unit: score on a scale] — Neurological functions are assessed by the Wolfram Unified Rating Scale (WURS). The WURS is divided into the following subscales: Physical Assessment and Behavioral Assessment. Physical Assessment (34 items rated on a scale from 0 = no symptoms to 4 = highest severity, minimum: 0, Maximum: 136) and Behavioral Assessment (9 items rated on frequency and severity from 0 = normal behavior to 3 = highest severity, Minimum: 0, Maximum: 27). Subscale scores are summed to calculate the total scores (minimum: 0, Maximum: 163). Higher total scores indicate more severe neurological manifestations.
  score on a scale | 21.3 (6.4) | 20.5 (2.8) | 20.8 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by Liver Function Tests
Description: The investigators assess the safety and tolerability of dantrolene sodium administered orally at upper end of therapeutic dose range for 6 months in patients with Wolfram syndrome. More specifically, the investigators perform liver function tests to check the levels of certain enzymes and proteins in participants' blood. Levels that are higher or lower than normal can indicate liver problems. The liver function tests include:
  Alanine transaminase (ALT), Aspartate transaminase (AST), Alkaline Phosphatase (AP), and bilirubin.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 8 | 11
Participants
  Baseline | 0 | 0
  6 months | 0 | 2

2. Secondary Outcome: Changes in C-peptide Levels in Participants Assessed by the ELISA Assay
Description: The investigators determine the effect of dantrolene sodium on residual beta cell functions. The investigators monitor base-line C-peptide levels in participants' blood. The investigators also monitor C-peptide levels in participant's blood during the oral mixed meal tolerance test. The night before the oral mixed meal tolerance test, the participants will turn their insulin pump basal rate to 50% of the normal rate at midnight or take half of their evening dose of Lantus insulin and fasted from midnight until the test at 8 a.m. The mixed meal consists of 6 ml/kg (maximum 360 ml) of Boost Original (Société des Produits Nestlé S.A., Vevey, Switzerland). Blood for glucose and C-peptide measurement will be drawn at time 0 (fasting) and 30 minutes after the Boost. If a subject's fasting glucose exceeds 11.1 mmol/l, the test will not be performed, but fasting glucose and C-peptide will be obtained.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 8 | 11
ng/mL
  Baseline | 0.34 (0.07) | 0.19 (0.05)
  6 months | 0.47 (0.13) | 0.30 (0.09)

3. Secondary Outcome: Changes in Visual Functioning in Participants Assessed by Visual Functioning Questionnaire-25.
Description: Changes in Visual Functioning in participants assessed by Visual Functioning Questionnaire-25.
  The Visual Functioning Questionnaire-25 (VFQ-25) is divided into several subdomains, each assessing a specific aspect of visual functioning and its impact on an individual's life. There are a total of 11 subdomains in the VFQ-25. To calculate the total score on the VFQ-25, we follow these steps:
  1. Calculate Subdomain Scores,
  2. Weighted Sum
  3. Calculate Total Score VFQ-25 provides scores that range from 0 to 100. The total score represents the overall impact of visual functioning on the individual's quality of life, with higher scores indicating better quality of life and less impact from vision problems.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 8 | 11
units on a scale
  Baseline | 68 (2.3) | 74.3 (1.3)
  6 months | 70.5 (2.9) | 73.5 (2.4)

4. Secondary Outcome: Changes in Best-corrected Visual Acuity in Participants Measured by LogMar Score
Description: Best-corrected visual acuity is assessed using the Snellen optotype and then converted into LogMar Scores (Minimum: -0.30, Maximum: 3.0). A higher LogMar score signifies poorer vision.
Time Frame: 6 months
Population: Patient 012 was excluded from analysis due to LogMar of 3 (No Light Perception)
Measure: Mean (Standard Error); unit: LogMAR
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 8 | 10
LogMAR
  Baseline | 0.6 (0.2) | 0.8 (0.2)
  6 months | 0.6 (0.2) | 0.9 (0.2)

5. Secondary Outcome: Changes in Neurological Functions in Participants Assessed by the Wolfram Unified Rating Scale (WURS)
Description: Neurological functions are assessed by the Wolfram Unified Rating Scale (WURS). The WURS is divided into the following subscales: Physical Assessment and Behavioral Assessment. Physical Assessment (34 items rated on a scale from 0 = no symptoms to 4 = highest severity, minimum: 0, Maximum: 136) and Behavioral Assessment (9 items rated on frequency and severity from 0 = normal behavior to 3 = highest severity, Minimum: 0, Maximum: 27). Subscale scores are summed to calculate the total scores (minimum: 0, Maximum: 163). Higher total scores indicate more severe neurological manifestations.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pediatric | Adult
Number analyzed (Participants) | 8 | 11
score on a scale
  Baseline | 21.3 (6.4) | 20.5 (2.8)
  6 months | 18.4 (5.7) | 18.6 (4.5)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Pediatric: Pediatric patients treated with dantrolene sodium
  dantrolene sodium: The purpose of this study is to assess the safety and tolerability of dantrolene sodium in patients with Wolfram syndrome. In addition, we will assess the efficacy of dantrolene sodium on the cardinal manifestations of Wolfram syndrome, including visual acuity, remaining beta cell functions, and neurological functions.
  There is a screening period up to 56 days, a 6-month treatment period and a 4-week safety follow-up period. Study assessments include medical & medication history, physical exams, neurological exams, eye exams, endocrine exams, vital signs, height, weight, electrocardiograms, blood and urine tests, pregnancy test if applicable, and questionnaires.
- Adult: Adult patients treated with dantrolene sodium
  dantrolene sodium: The purpose of this study is to assess the safety and tolerability of dantrolene sodium in patients with Wolfram syndrome. In addition, we will assess the efficacy of dantrolene sodium on the cardinal manifestations of Wolfram syndrome, including visual acuity, remaining beta cell functions, and neurological functions.
  There is a screening period up to 56 days, a 6-month treatment period, and a 4-week safety follow-up period. Study assessments include medical & medication history, physical exams, neurological exams, eye exams, endocrine exams, vital signs, height, weight, electrocardiograms, blood and urine tests, pregnancy test if applicable, and questionnaires.
Arm/Group | Pediatric | Adult
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 8/8 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric (N=8) | Adult (N=11)
Diarrhea (Gastrointestinal disorders) | 2 | 3
Weakness (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 1
Elevated Hepatic enzymes (Hepatobiliary disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Gastrointestinal upset (Gastrointestinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Hypoglycemia (mild) (Endocrine disorders) | 3 | 4
Headaches (Nervous system disorders) | 2 | 4
hyponatremia (Renal and urinary disorders) | 1 | 3
Hyperglycemia (Endocrine disorders) | 2 | 1
Urinary Tract Infection (Renal and urinary disorders) | 1 | 3
Hyperkalemia (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinovirus infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Knee Infection (Infections and infestations) | 1 | 0
Tics (Nervous system disorders) | 1 | 0
Knee Effusions (Skin and subcutaneous tissue disorders) | 1 | 0
Hit by car (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (Nervous system disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02829268/Prot_SAP_000.pdf